CLINICAL TRIAL: NCT06011772
Title: A Phase 0 Study of EGF-Depleting Therapy CIMAvax-EGF in Combination With Standard Therapy for RAS- and BRAF Wild-Type Metastatic Colorectal Cancer
Brief Title: EGF-Depleting Therapy CIMAvax-EGF in Combination With Standard Therapy for RAS- and BRAF Wild-Type Metastatic Colorectal Cancer
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I 1578122
Record Dates: First submitted 2023-08-21; First posted 2023-08-25 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Colo-rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — CIMAvax EGF; Epidermal Growth Factor; Vaccines; Leucovorin; Oxaliplatin; Fluorouracil; Bevacizumab; Irinotecan; Cetuximab; Metastasectomy; Panitumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Cohort A (Experimental): LOADING PHASE: Patients receive CIMAvax-EGF IM on days 1 and 15. Treatment repeats every 28 days for 2 cycles in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE PHASE: Patients receive CIMAvax-EGF IM on day 15. Treatment repeats every 28 days for 10 cycles in the absence of disease progression or unacceptable toxicity. Patients also receive chemotherapy consisting of leucovorin IV, oxaliplatin IV over 2 hours, and fluorouracil IV and bevacizumab IV over 10 minutes on days 1 and 15. Treatment repeats every 2 weeks for 10 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo collection of blood samples throughout the trial.
  Interventions: Biological: Recombinant Human EGF-rP64K/Montanide ISA 51 Vaccine; Drug: Leucovorin; Drug: Oxaliplatin; Drug: Fluorouracil; Biological: Bevacizumab; Drug: Irinotecan; Biological: Cetuximab; Procedure: Biospecimen collection; Procedure: Computed Tomography; Biological: Panitumumbab
- Cohort B (Experimental): LOADING PHASE: Patients receive CIMAvax-EGF IM on days 1 and 15. Treatment repeats every 28 days for 2 cycles in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE PHASE: Patients receive CIMAvax-EGF IM on day 15. Treatment repeats every 28 days for 10 cycles in the absence of disease progression or unacceptable toxicity. Patients also receive FOLFIRI consisting of irinotecan IV, leucovorin IV over 90 minutes, and fluorouracil IV and cetuximab IV over 120 minutes on days 1 and 15. Treatment repeats every 2 weeks for 10 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo collection of blood samples throughout the trial.
  Interventions: Biological: Recombinant Human EGF-rP64K/Montanide ISA 51 Vaccine; Drug: Leucovorin; Drug: Oxaliplatin; Drug: Fluorouracil; Biological: Bevacizumab; Drug: Irinotecan; Biological: Cetuximab; Procedure: Biospecimen collection; Procedure: Computed Tomography; Biological: Panitumumbab
- Cohort C (Experimental): Description LOADING PHASE: Patients receive CIMAvax-EGF IM on days 1 and 15. Treatment repeats every 28 days for 2 cycles in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE PHASE: Patients receive CIMAvax-EGF IM on day 15. Treatment repeats every 28 days for 10 cycles in the absence of disease progression or unacceptable toxicity. Patients also receive mFOLFOX6 and cetuximab, FOLFOX6 and bevacizumab, or mFOLFOX6 per investigators preference. Treatment repeats every 2 weeks for 10 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo metastasectomy 4-8 weeks after first maintenance phase dose. Patients undergo collection of blood samples throughout the trial.
  Interventions: Biological: Recombinant Human EGF-rP64K/Montanide ISA 51 Vaccine; Drug: Leucovorin; Biological: Bevacizumab; Biological: Cetuximab; Procedure: Metastasectomy; Procedure: Biospecimen collection

INTERVENTIONS:
Biological: Recombinant Human EGF-rP64K/Montanide ISA 51 Vaccine — Given IM
  Other Names: Cimavax; CIMAvax EGF; Epidermal Growth Factor (EGF) Vaccine
Drug: Leucovorin — Given IV
Drug: Oxaliplatin — Given IV
  Arms: Cohort A; Cohort B
Drug: Fluorouracil — Given IV
  Arms: Cohort A; Cohort B
Biological: Bevacizumab — Given IV
Drug: Irinotecan — Given IV
  Arms: Cohort A; Cohort B
Biological: Cetuximab — Given IV
Procedure: Metastasectomy — Undergo metastasectomy
  Arms: Cohort C
Procedure: Biospecimen collection — Undergo collection of blood samples
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT SCAN
  Arms: Cohort A; Cohort B
Biological: Panitumumbab — Given IV
  Other Names: ABX-EGF; ABX-EGF Monoclonal Antibody
  Arms: Cohort A; Cohort B

SUMMARY:
The purpose of this study is to determine the immunogenicity of the CIMAvaxEGF® vaccine (that is, its effectiveness in inducing an anti-tumor immune response) in patients with metastatic KRAS/NRAS/BRAF wild-type gene colorectal cancer, when given in combination with standard therapies used in the treatment of advanced colorectal cancer.

DETAILED DESCRIPTION:
Primary Objective

- Determine the immunogenicity of CIMAvax in patients with metastatic, KRAS/NRAS/BRAF wild type CRC in combination with Chemotherapy plus appropriate biologic agent in 1st or 2nd/3rd line setting and chemotherapy plus anti-EGFR therapy in 2nd/3rd line setting.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed metastatic adenocarcinoma of colon or rectum that cannot be removed by surgery without prior systemic therapy for advanced disease (prior adjuvant chemotherapy completed >12 months from diagnosis of metastatic or advanced disease is allowed) for cohorts A and C and with one prior line of therapy but no more than 2 prior lines of therapy for advanced disease (prior adjuvant chemotherapy completed <12 months from diagnosis of metastatic or advanced disease is considered one line of therapy).

  * Cohort A: May have received 1 cycle of chemotherapy± appropriate biologic agent pending results of RAS and BRAF. If results determine patient is eligible, the patient will be enrolled and will receive the addition of CIMAvax + Bevacizumab or CIMAvax+ anti-EGFR therapy in their second cycle.
  * Cohort B: Patients with RAS- and BRAF wild-type metastatic CRC who have received at least one but no more than 2 prior therapies for advanced disease
  * Cohort C: Patients with RAS- and BRAF wild-type metastatic CRC who have not received prior therapy for advanced disease and are candidates for metastatic disease resistant resection (one cycle of standard chemotherapy with or without appropriate biologic agent is allowed)
* KRAS/NRAS/BRAF wild-type.
* Have an ECOG Performance Status of 0-2
* Patients must have adequate organ and marrow function as defined below:

  * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
  * Platelets ≥ 75 x 10^9/L
  * Hemoglobin ≥ 8 g/dL
  * Creatinine clearance> 60 mL/min (Cockcroft-Gault Equation)
  * ALT and AST ≤ 3 x ULN (ALT and AST ≤ 5 x ULN is acceptable if liver metastases are present
  * Total bilirubin ≤ 1.5x ULN. For patients with well documented Gilbert's syndrome, total bilirubin ≤ 3x ULN with direct bilirubin within normal range
* Have measurable disease per RECIST 1.1 criteria present.
* Participants of child-bearing potential must agree to use adequate contraceptive methods (e.g., hormonal or barrier method of birth control; abstinence) prior to study entry. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Participant must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure.
* Participant agrees to provide paired-tumor biopsy tissue while on study (cohort A and B) or allow tissue to be taken during surgery (cohort C)

Exclusion Criteria:

* Toxicity ≥Grade 2 from prior chemotherapy with exception to Grade 2 peripheral neuropathy..
* Other cancer requiring active treatment.
* Prior exposure to anti-EGFR monoclonal antibody (i.e. cetuximab or panitumumab) for colorectal cancer treatment is exclusionary to Cohort A and C only
* Participants with Her2 positive mutational status
* Had major surgery within 4 weeks prior to starting study drug or has not recovered from major side effects (tumor biopsy is not considered major surgery) resulting from a prior surgery.
* Has known immunosuppressive disease (e.g. HIV, AIDS or other immune depressing disease). Testing is not mandatory.
* Participants with known active brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* Active, clinically serious infections or other serious uncontrolled medical conditions or psychiatric illness/social situations that would limit compliance with study requirements.
* History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, or is not in the best interest of the patient to participate, in the opinion of the treating Investigator, including, but not limited to:

  * Myocardial infarction or arterial thromboembolic events within 6 months prior to baseline or severe or unstable angina, New York Heart Association (NYHA) Class III or IV disease
  * History of documented congestive heart failure (New York Heart Association functional classification III or IV) within 6 months prior to baseline
  * Uncontrolled hypertension (SBP>160/DBP>100 despite medical intervention).
  * History of myocarditis of any etiology
  * History of ventricular arrhythmias
* Active major or clinically significant bleeding based on the International Society on Thrombosis and Hemostasis definition.
* Pregnant or nursing female participants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2023-12-18 (Actual); Primary Completion 2025-07-05 (Actual); Study Completion 2026-12-04 (Estimated)

PRIMARY OUTCOMES:
Immunogencity of vaccine | up to 60 days after last dose
  Percentage of patients with antibody titers greater than or equal to 1:4000 using a 90% confidence interval obtained by Jeffery's prior method

SECONDARY OUTCOMES:
Progression free survival | time from treatment until disease progression, death or last follow up assesed up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Deepak Vadehra, Principal Investigator — Roswell Park Comprehensive Cancer Center
Locations (1):
- Roswell Park Comprehensive Cancer Center, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No